CLINICAL TRIAL: NCT05829408
Title: KOPPeling: Help From Your Own Circle
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Collaborators: Accare (Other); WIJ Groningen (Unknown); GGZ Friesland (Other); Amaryllis Leeuwarden (Unknown); Hanzehogeschool Groningen (Unknown); Lentis (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 10196
Record Dates: First submitted 2023-02-21; First posted 2023-04-25 (Actual); Last update posted 2024-08-01 (Actual); Status verified 2024-07

CONDITIONS: Children of Parents With a Mental Illness (COPMI)
Keywords: COPMI; Prevention; Social participation; Mental illness
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (KOPPeling) (Other): In this arm participants directly receive the KOPPeling intervention.
  Interventions: Behavioral: KOPPeling
- Waiting list (Other): In this arm participants are placed on a waiting list (ten to twelve weeks) before receiving the KOPPeling intervention.
  Interventions: Behavioral: KOPPeling

INTERVENTIONS:
Behavioral: KOPPeling — KOPPeling lasts ten to twelve weeks and will be administered by health care professionals.

SUMMARY:
The goal of this randomized clinical trial is to test the effectiveness of the KOPPeling intervention that aims at unburdening COPMI (Children Of Parents with a Mental Illness). COPMI are at risk of overtaking the tasks of their parents when their parents are unable to fulfil such due to their psychiatric condition. By overtaking tasks and the urge to always take care of their parents, COPMI often do not participate in outdoor activities, which are necessary for their socio-emotional development. Moreover, insufficient socio-emotional development and parentification are risk factors for the development of psychiatric conditions.

KOPPeling is an intervention for COPMI families that focuses on activating the social networks of the families. Within KOPPeling, a strategic plan will be developed and carried out with the goal of receiving support from the social network that will overtake tasks of the family to unburden COPMI.

This study aims to answer the following questions:

1. To what extent does KOPPeling lead to an increase in Quality of Life (QoL) among COPMI?
2. To what extent does KOPPeling lead to an increase in mental health among COPMI?
3. To what extent does KOPPeling lead to a reduction of parenting stress among COPMI parents?
4. To what extent does KOPPeling lead to an increase in outdoor activities among COPMI?
5. How does KOPPeling affect the feelings of guilt of COPMI when engaging in outdoor activities?
6. What pre-conditions are needed to make KOPPeling widely applicable?
7. What are the long-term effects of KOPPeling on the QoL and psychological problems among COPMI and parental stress among COPMI parents?

Participants will participate in the ten-to-twelve-week long KOPPeling intervention. Researchers will compare the intervention group with a waiting list control group to test the effect of KOPPeling on the QoL and mental health of COPMI and parental stress of parents.

ELIGIBILITY:
Inclusion Criteria:

* The family has children aged 0-18 living at home
* The parental disorder influences the parent's (or parents') ability to carry out several important parental tasks, placing their offspring at risk of taking over these tasks

Exclusion Criteria:

- The family has no existing social network

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-04-23 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Change in Quality of Life (QoL) of COPMI | At T0 (baseline, start of intervention), T1 (end of intervention) and T2 (three months after the end of intervention), total time frame: 22 to 24 weeks
  QoL of COPMI, which will be assessed with the KIDSCREEN-27. The KIDSCREEN-27 includes 27 items measuring five dimensions of QoL on a Rasch scale including: 1) physical well-being, 2) psychological well-being, 3) autonomy and parent relation, 4) peers and social support, and 5) school environments. Each item is measured on a five-point Likert scale. Some items are negatively formulated through which the item scores need to be reversed. The overall score is calculated by summing up all the items. Therefore, higher scores indicate higher QoL.

SECONDARY OUTCOMES:
Change in mental health of COPMI | At T0 (baseline, start of intervention), T1 (end of intervention) and T2 (three months after the end of intervention), total time frame: 22 to 24 weeks
  The mental health of COPMI, which will be assessed with the Strengths and Difficulties Questionnaire (SDQ). The SDQ consists out of 25 items (five scales of five items each) including the following subscales: 1) emotional symptoms, 2) conduct problems, 3) hyperactivity/inattention, 4) peer relationships problem and 5) prosocial behaviour.
  Each attribute is scored on a zero to ten scale. While a score of 0 is the best outcome concerning the emotional, conduct, hyperactivity, and peer relationship scale (adding up to a 0 to 40 scale), a score of 10 is the best outcome concerning the pro-social behaviour scale.
Change in parental stress of COPMI parents | At T0 (baseline, start of intervention), T1 (end of intervention) and T2 (three months after the end of intervention), total time frame: 22 to 24 weeks
  The parental stress of COPMI parents, which will be assessed with the Nijmeegse Ouderlijke Stress Index (NOSI-K). The NOSI-K includes 25-items assessing parental perceived difficulty in child rearing. Each item, which states a parental-stress-related statement, is rated on a five-point Likert scale ranging from 1 (totally disagree) to (totally agree).
Change in engagement in outdoor activities of COPMI | For one week after the start of the intervention and one week before the end of the intervention
  The engagement in outdoor activities will be measured in an ecological momentary assessment.
Change in guilt of COPMI when engaging in outdoor activities | For one week after the start of the intervention and one week before the end of the intervention
  The associated guilt of engaging in outdoor activities of COPMI will be assessed in an ecological momentary assessment in which the Guilt and Shame Questionnaire for Adolescents of Parents with a Mental Illness (GSQ-APMI) will be used. The GSQ-APMI includes 10 items. Five items were developed to measure shame and five items to measure guilt. A total score is not applicable as the GSQ-APMI results in two scores: one reflecting feelings of guilt and one reflecting feelings of shame. Higher scores reflect greater feelings of guilt or shame.
Experiences of the social networks made with KOPPeling | At the end of the intervention (ten to twelve weeks after the start of the intervention)
  The experiences of the social network with KOPPeling, which will be assessed in a qualitative interview with a purposive sample taken from the social networks of included families.
Promoting and hindering factors of making KOPPeling a widely applicable intervention | At the end of the intervention (ten to twelve weeks after the start of the intervention)
  The promoting and hindering factors for making the intervention widely applicable, which will be assessed with the Measuring Instrument for Determinants of Innovations (MIDI).

CONTACTS AND LOCATIONS:
Overall Officials: Frederike Jörg, Dr., Principal Investigator — University Medical Center Groningen
Locations (1):
- UMC Groningen, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravens-Sieberer U, Gosch A, Rajmil L, Erhart M, Bruil J, Duer W, Auquier P, Power M, Abel T, Czemy L, Mazur J, Czimbalmos A, Tountas Y, Hagquist C, Kilroe J, Kidscreen Group E. KIDSCREEN-52 quality-of-life measure for children and adolescents. Expert Rev Pharmacoecon Outcomes Res. 2005 Jun;5(3):353-64. doi: 10.1586/14737167.5.3.353. PMID 19807604
- [Background] Muris P, Meesters C, van den Berg F. The Strengths and Difficulties Questionnaire (SDQ)--further evidence for its reliability and validity in a community sample of Dutch children and adolescents. Eur Child Adolesc Psychiatry. 2003 Jan;12(1):1-8. doi: 10.1007/s00787-003-0298-2. PMID 12601558
- [Background] van Widenfelt BM, Goedhart AW, Treffers PD, Goodman R. Dutch version of the Strengths and Difficulties Questionnaire (SDQ). Eur Child Adolesc Psychiatry. 2003 Dec;12(6):281-9. doi: 10.1007/s00787-003-0341-3. PMID 14689260
- [Background] Shiffman S, Stone AA, Hufford MR. Ecological momentary assessment. Annu Rev Clin Psychol. 2008;4:1-32. doi: 10.1146/annurev.clinpsy.3.022806.091415. PMID 18509902
- [Background] Fleuren MA, Paulussen TG, Van Dommelen P, Van Buuren S. Towards a measurement instrument for determinants of innovations. Int J Qual Health Care. 2014 Oct;26(5):501-10. doi: 10.1093/intqhc/mzu060. Epub 2014 Jun 20. PMID 24951511